CLINICAL TRIAL: NCT03344926
Title: ACTsmart - Feasibility of Smart Phone Delivered ACT Treatment for Adults With Longstanding Pain
Brief Title: Smart Phone ACT Treatment for Adults With Longstanding Pain - a Pilot Study
Acronym: ACTsmart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rikard Wicksell (Other)
Collaborators: AFA Insurance (Industry)
Responsible Party: Sponsor-Investigator, Rikard Wicksell, Associate professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1638-31/2:2
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain
Keywords: Acceptance and Commitment therapy; ACT; CBT; Smart phone; Internet; Intervention
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Pilot study of treatment delivery in a new format.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACTsmart (Experimental): ACT treatment via a smart phone application
  Interventions: Behavioral: ACTsmart

INTERVENTIONS:
Behavioral: ACTsmart — Participant receive ACT treatment via a smart phone application, including psychologist support via a message function within the application.
  Treatment content is divided into four modules:
  1. education about pain behaviors, exposure and acceptance and commitment therapy
  2. education about pain physiology
  3. exercises on changing behaviors, acceptance, mindfulness, defusion and exposure
  4. value based exposure in the participant's daily life

SUMMARY:
The aims are to test feasibility and preliminary effects of a smart phone delivered ACT treatment for adults with longstanding pain.

The hypotheses are that

1. ACTsmart will be a feasible and accessable treatment delivery form
2. ACTsmart will improve function and quality of life

DETAILED DESCRIPTION:
Chronic pain affects 12-30% of the population and often results in depression, disability, and reduced daily function and quality of life. Medical strategies are often ineffective or insufficient to alleviate symptoms and increase functioning. Instead, the empirical support for cognitive behavior therapy (CBT) is today well established, and such interventions are commonly seen as critically important for patients with chronic pain. However, modest effects sizes calls for further improvements. Recent developments within CBT, particularly Acceptance and Commitment Therapy (ACT), have suggested the utility of acceptance and mindfulness strategies to manage pain and distress. The body of evidence for ACT has grown rapidly during the past decade, and ACT is today listed by the American Psychological Association as a treatment for chronic pain, with strong empirical support.

Internet-delivered ACT Despite the increased empirical support for ACT the availability is still very limited, and a large number of patients do not receive this treatment. In other domains, the accessibility of empirically supported treatments has increased during the past decade due to the development of methods to deliver the treatment via internet. For example, a large number of studies illustrate the utility of internet-delivered CBT for anxiety, insomnia and depression, with treatment effects similar to those obtained in studies with face-to-face treatment. Few studies have yet evaluated internet-delivered ACT (iACT) for chronic pain, but a recent pilot study from our group with participants suffering from fibromyalgia (n=41) illustrated very promising results that warrant further studies to evaluate the effects of this treatment.

To make treatment more accessible and present in patients' daily life we will use a smart phone application to deliver treatment.

Recruitment Patients will be recruited through self referral. Information regarding the study will be provided through newspapers and social media, as well as in direct communication with pain clinics and primary care units, including instructions regarding e.g. eligibility and how to sign up. Once patients have been found eligible and expressed interest in study participation they will be assessed by a psychologist, and when needed by a pain physician, via semi-structured interviews to confirm eligibility and to ensure that the patient meet the study criteria. Informed consent is obtained from all participants prior to the assessment.

Statistical methods Evaluations of treatment effects are primarily based on intent-to-treat analyses. The statistical approach will primarily be based on linear multilevel modeling (LMM), which takes into account dependencies between repeated measures and differences between patients in pre-treatment status and treatment response (i.e. random effects modeling) and also provide means of handling missing data. More traditional methods, such as ANOVA and hierarchical regression, may also be utilized when appropriate.

Interviews Evaluations of feasibility and as a base for further development of the smart phone application will be done via semi structured interviews during and after treatment period.

ELIGIBILITY:
Inclusion Criteria:

* a pain duration of ≥ 6 months;
* able to read and write in Swedish
* have access to a smart phone with internet access
* no planned changes in medication use, or any other changes in interventions for their pain planned

Exclusion Criteria:

* injury or illness that require immediate assessment or different treatment, or that is expected to progress significantly during the next 6 months
* unstable medication (planned changes in medication during next 4 months)
* ACT or CBT treatment during the past 3 months
* severe psychiatric co-morbidity (e.g. high risk of suicide) as assessed by the psychologist in a semi-structured interview

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Pain Interference Index (changes between assessments) | Baseline, 8 weekly ratings, post (8 weeks), follow ups three, six and twelve months post treatment
  Self rated measure of daily functioning related to pain

SECONDARY OUTCOMES:
Psychological Inflexibility in Pain Scale (changes) | Baseline, 8 weekly ratings, post (8 weeks), follow ups three, six and twelve months post treatment
  Self rated psychological inflexibility related to pain. Total score min 12, max 84, lower values are interpreted as higher psychological flexibility, higher values interpreted as lower psychological flexibility. Two subscales; fusion (4-28) and avoidance (8-56) are summed to compute a total score.
Valuing Questionnaire (changes) | Baseline, 8 weekly ratings, post (8 weeks), follow ups three, six and twelve months post treatment
  Self rated progress and obstacles in valued actions. The Valuing Questionnaire consists of two subscales: progress (0-30) och obstacles (0-30). No total score is computed. On the obstacle subscale higher scores are worse, and on the progress subscale higher scores are better.
Patient Health Questionnaire 9 (changes) | Baseline, post (8 weeks), follow ups three, six and twelve months post treatment
  Self rated depressive symptoms. Score is summed to a possible range of 0 to 27. Higher scores are interpreted as worse.
European Quality of Life Five Dimensions Questionnaire (changes) | Baseline, post (8 weeks), follow ups three, six and twelve months post treatment
  Self rated quality of life. Scores are calculated to a number between 0 and 1, where 0 in theory is equal to death, and 1 is considered equal to perfect quality of life.
Insomnia Severity Index (changes) | Baseline, post (8 weeks), follow ups three, six and twelve months post treatment
  Self rated degree of insomnia
Pain intensity (changes) | Baseline, post (8 weeks), follow ups three, six and twelve months post treatment
  Self rated degree of pain during last week on a scale from 0-10
Occupational status (changes) | Baseline, post (8 weeks), follow ups three, six and twelve months post treatment
  Self reported occupational status indicated on a pre specified list, including sick leave and/or sick retirement
Generalized Anxiety Disorder - 7 (changes) | Baseline, post (8 weeks), follow ups three, six and twelve months post treatment
  Self rated symptoms of anxiety
Medication use (changes) | Baseline, post (8 weeks), follow ups three, six and twelve months post treatment
  Self reported medicine use

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Wicksell, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gentili C, Zetterqvist V, Rickardsson J, Holmstrom L, Ljotsson B, Wicksell R. Examining predictors of treatment effect in digital Acceptance and Commitment Therapy for chronic pain. Cogn Behav Ther. 2023 Jul;52(4):380-396. doi: 10.1080/16506073.2023.2191826. Epub 2023 Mar 27. PMID 36971108